CLINICAL TRIAL: NCT03864172
Title: Effects of Soluble Corn Fiber on BMC, BMD and Bone Biomarkers of Pre-pubertal Boys and Girls : a Randomized Controlled Trial
Brief Title: Soluble Corn Fiber on BMD in Pre-pubertal Boys and Girls (PREBONE-Kids)
Acronym: PREBONE-Kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMU University, Malaysia (Other)
Collaborators: Tate & Lyle (Industry)
Responsible Party: Principal Investigator, Winnie Chee, Principal Investigator, IMU University, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: InternationalMU
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Bone Health

STUDY DESIGN:
Intervention Model Description: Randomised controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual intake + placebo fruit juice (Placebo Comparator): Placebo fruit flavoured juice powder
  Interventions: Dietary Supplement: Usual intake + placebo fruit juice
- Usual intake +SCF fruit juice (Active Comparator): Fruit flavoured juice powder added with 12 g soluble corn fiber (SCF)
  Interventions: Dietary Supplement: Usual intake+SCF fruit juice
- Adequate calcium +fruit juice placebo (Active Comparator): Placebo fruit flavoured juice powder added with 600 mg calcium to meet RNI intake
  Interventions: Dietary Supplement: Adequate calcium + placebo fruit juice
- Adequate calcium + SCF fruit juice (Active Comparator): Fruit flavoured juice powder added with 12 g soluble corn fiber (SCF) and 600 mg calcium to meet RNI intake
  Interventions: Dietary Supplement: Adequate calcium+ SCF fruit juice

INTERVENTIONS:
Dietary Supplement: Usual intake + placebo fruit juice — Participants will consume 200 mls of placebo fruit flavoured juice
  Arms: Usual intake + placebo fruit juice
Dietary Supplement: Usual intake+SCF fruit juice — Participants will consume 200 mls of fruit flavoured juice containing 12 g soluble corn fiber (SCF)
  Arms: Usual intake +SCF fruit juice
Dietary Supplement: Adequate calcium + placebo fruit juice — Participants will consume 200 mls of placebo fruit flavoured juice added with 600 mg calcium to meet RNI
  Arms: Adequate calcium +fruit juice placebo
Dietary Supplement: Adequate calcium+ SCF fruit juice — Participants will consume 200 mls of fruit flavoured juice containing 12 g soluble corn fiber (SCF) added with 600 mg calcium to meet RNI
  Arms: Adequate calcium + SCF fruit juice

SUMMARY:
The aim of this study is to investigate the effects of soluble corn fiber (SCF) on bone mineral content (BMC) and bone mineral density (BMD) in pre-pubertal boys and girls. The hypothesis to be tested is: SCF will lead to greater increase of BMD, as measured with densitometry in both low calcium as well as high calcium intakes compared to placebo.

DETAILED DESCRIPTION:
Main objective To investigate the effects of soluble corn fiber (SCF) supplementation on bone mineral content (BMC) and bone mineral density (BMD) in pre-pubertal boys and girls.

Secondary objectives

The secondary objectives are:

To investigate changes in bone formation and bone resorption markers in response to soluble corn fiber supplementation in the diet of prepubertal boys and girls consuming adequate calcium intake vs placebo To investigate changes in body composition in response to soluble corn fiber supplementation in the diet of prepubertal boys and girls consuming adequate calcium intake vs placebo

Hypothesis Soluble corn fiber would lead to improved BMC and BMD accrual in pre-pubertal children compared to placebo.

Study design The proposed study is a double blind, randomized, single center, parallel design trial

Duration of study The duration of the study intervention would be 12 months

ELIGIBILITY:
Inclusion Criteria

* Screened to be generally healthy as determined by standard medical assessment on physical and mental health
* Tanner stage 2 based on breast development for girls, and pubic hair in boys. Girls will have to be premenarcheal
* Having obtained his/her informed consent and parents or legal guardians consent

Exclusion Criteria:

* History of serious medical conditions such as intestinal or severe metabolic diseases, disorders such as diabetes, renal, hepatic or pancreatic diseases, disorders, ulcer, hyperthyroidism, malignance, chronic malnutrition, anaemia
* History or on therapy with medication known to interfere with bone metabolism such as steroids, hormones, diuretics, cortisone or anti-seizure medication
* Taking regularly any nutritional supplements and unwilling to stop for the study

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 243 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Bone mineral density ( BMD) | 12 months
  BMD at total body and lumbar spine L1-L4
Bone mineral content (BMC) | 12 months
  BMC at total body and lumbar spine L1-L4

SECONDARY OUTCOMES:
Bone biomarkers | 12 months
  Serum CTX1, P1NP, osteocalcin & BAP

CONTACTS AND LOCATIONS:
Overall Officials: Winnie SS Chee, PhD, Principal Investigator — IMU University, Malaysia
Locations (1):
- International Medical University, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arasu K, Chang CY, Wong SY, Ong SH, Yang WY, Chong MHZ, Mavinkurve M, Khoo EJ, Chinna K, Weaver CM, Chee WSS. Effect of soluble corn fibre and calcium supplementation on bone mineral content and bone mineral density in preadolescent Malaysian children-a double-blind randomised controlled trial (PREBONE-Kids Study). Osteoporos Int. 2023 Apr;34(4):783-792. doi: 10.1007/s00198-023-06702-0. Epub 2023 Feb 21. PMID 36808216